CLINICAL TRIAL: NCT05839756
Title: Predicting Post Extubation Stridor in Patients With Intermaxillary Fixation
Brief Title: Predicting Post Extubation Stridor After Maxillomandibular Fixation
Acronym: airway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Post Extubation Stridor
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Stridor; Larynx Edema
MeSH Terms: conditions — Respiratory Sounds; Laryngeal Edema | interventions — Budesonide; Saline Solution

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated into two equal groups via opaque coded envelopes
Who Masked: Participant, Investigator
Masking Description: The preoperative aerosolized drug will be applied by an anesthetist who is not involved in further patient care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (C) group (Placebo Comparator): normal saline will be nebulized
  Interventions: Drug: normal saline
- Budesonide (B) group (Active Comparator): budesonide will be nebulized
  Interventions: Drug: budesonide

INTERVENTIONS:
Drug: budesonide — 2 ml nebulized budesonide (containing 1 mg) diluted in 3 ml of normal saline will be nebulized preoperatively
  Arms: Budesonide (B) group
Drug: normal saline — 5 ml normal saline will be nebulized preoperatively
  Arms: control (C) group

SUMMARY:
Endotracheal intubation can induce laryngotracheal injury which results in narrowing of the airway due to edema of the glottis. This can increase the risk of development of post-extubation stridor (PES)

DETAILED DESCRIPTION:
Ultrasound (US) is a useful and non-invasive tool for the evaluation of vocal cords and laryngeal morphology in intubated patients. The laryngeal air-column width (LACW), Laryngeal air column width difference (LACWD), and laryngeal air-column width ratio (LACWR) measured by ultrasound can potentially identify patients at risk of post-extubation stridor, in whom caution should be taken after extubation.

The cuff-leak test can predict successful extubation through using the difference between the expired tidal volume with the cuff inflated and with the cuff deflated; the higher the leak, the lower the likelihood that post-extubation stridor will occur.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* American Society of Anesthesiologists status I and II
* undergoing elective maxillomandibular fixation surgeries under general anesthesia with nasal endotracheal intubation

Exclusion Criteria:

* patients' refusal
* pregnant females
* patients with body mass index <18.5 or ≥ 35 kg/m2
* risk of aspiration
* cardiorespiratory disorder
* neuromuscular disease
* uncontrolled diabetes mellitus
* gastrointestinal bleeding
* on chronic steroid therapy
* intubated patients or were intubated or had upper airway infection within 1 week prior to surgery
* history of any pathology, radiotherapy or surgery in the neck
* had difficult laryngeal US plane (as neck wound)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2025-02-25 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Laryngeal air column width ratio | immediately before extubation

SECONDARY OUTCOMES:
The duration of nasal endotracheal intubation | Procedure (from nasal endotracheal intubation till extubation)
  min
endotracheal tube insertion depth | immediately after intubation
  cm
The incidence of epistasis occurrence during nasotracheal intubation | immediately after intubation
  4-point verbal descriptor scale (0=no symptoms, 1=mild, 2=moderate, 3=severe)
Expiratory tidal volume immediate after intubation with the cuff inflated | immediately after intubation
  ml

OTHER OUTCOMES:
Expiratory tidal volume immediate after intubation with the cuff deflated | immediately after intubation
  ml
Expiratory tidal volume immediate before extubation with the cuff inflated | immediately before extubation
  ml
Expiratory tidal volume immediate before extubation with the cuff deflated | immediately before extubation
  ml
cuff leak volume | immediate after intubation and immediate before extubation
  ml
Laryngeal air column width | before intubation
  mm
Laryngeal air column width | immediate after intubation during the balloon-cuff inflation and during balloon-cuff deflation
  mm
Laryngeal air column width | immediate before extubation during the balloon-cuff inflation and during balloon-cuff deflation
  mm
Laryngeal air column width difference | immediate after intubation and immediate before extubation
  mm
incidence of postoperative sore throat, dysphonia, swallowing disorders or PES. | First postoperative day
  4-point verbal descriptor scale (0=no symptoms, 1=mild, 2=moderate, 3=severe)

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Ahmed AboZeid, Al Mansurah, Egypt